CLINICAL TRIAL: NCT01769820
Title: Developmental Clinical Studies - Reversing Endometrial Glucocorticoid Deficiency in Heavy Menstrual Bleeding
Brief Title: Dexamethasone for Excessive Menstruation
Acronym: dexFEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Hilary Critchley, Professor of Reproductive Medicine, University of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: dexfemv2
Record Dates: First submitted 2012-12-19; First posted 2013-01-17 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Heavy Menstrual Bleeding
Keywords: Heavy menstrual bleeding (HMB); Dexamethasone; glucocorticoid
MeSH Terms: conditions — Menorrhagia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): Study 1, and study2(2 arms); Dexamethasone 1.5mg daily Study 3 (adaptive -7 arms): Dexamethasone of 0.4, 0.8, 1.0, 1.2, 1.5, and 1.8 mg total dose per day
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dexamethasone — studies 1&2:0.75mg twice daily for 5 days, starting on day LH (Luteinising Hormone)+8 of menstrual cycle; Study 3 (adaptive) 0.2,0.4,0.5,0.75,0.8,0.9mg twice daily as above
  Other Names: D07AB19
  Arms: Dexamethasone
Drug: placebo
  Arms: Placebo

SUMMARY:
This study builds on previous research which has provided compelling evidence that deficient activity of glucocorticoids in the endometrium is a cause of increased menstrual bleeding. This study aims to demonstrate that a glucocorticoid (dexamethasone), already in common use for other conditions, (eg to treat medical conditions such as asthma and rheumatoid arthritis in early pregnancy), will reverse the endometrial glucocorticoid deficiency and as a result reduce menstrual blood loss.

The study is in two stages, a 12 month workup stage and a 3 year, response adaptive, dose-finding randomised controlled trial. The first stage involves two workup clinical studies to gather preliminary safety and efficacy data from first-in-Heavy Menstrual Bleeding use of oral dexamethasone. They will also provide methodological data for a series of simulation studies to determine a robust adaptive trial design specification.

Workup study 1: is unblinded, six patients will be given Dexamethasone (0.75mg twice daily) for 5 days during two consecutive menstrual cycles and will have an endometrial biopsy and MRI on two occasions (in a nontreated cycle, and the second of the cycles treated with Dexamethasone). Workup study 2; is a doubleblind crossover trial of 14 women -2 treatment blocks of two cycles each, with either placebo or Dexamethasone (0.75mg twice daily), randomised to order of treatments blocks - placebo then Dexamethasone, or vice-versa.

Adaptive trial: 54 month double-blind, placebo controlled trial of 108 women to evaluate the effect of Dexamethasone across a range of doses with the aim of identifying the optimal dose to be studied in a subsequent Phase III trial.

Participants will be randomised to receive one of 6 active doses or placebo over 3 menstrual cycles.

All studies will involve asking participants to complete menstrual diaries and to carry out menstrual blood loss collections to objectively measure blood loss.

The investigators' proposed approach is novel use of synthetic glucocorticoid to "rescue" luteal phase deficiency of cortisol, and thus improve endometrial vasculature and hence vasoconstriction when menses commences, and thus reduce menstrual bleeding.

DETAILED DESCRIPTION:
Background Menstrual bleeding complaints affect quality of life and comprise a substantial societal burden, including major impact on health care use and costs. Current medical therapy for heavy menstrual bleeding (HMB) is often ineffective and/or associated with unacceptable side effects. There is unmet clinical need for targeted, effective, medical treatment strategies for HMB. The investigators' findings from research into mechanisms in HMB has led to the conclusion that women with HMB have enhanced endometrial inactivation of cortisol by 11βHSD2 resulting in local endometrial glucocorticoid deficiency, changes in prostaglandin (PG) production, and altered structure and deficient vasoconstriction of the endometrial vasculature. The investigators therefore anticipate that luteal phase "rescue" of endometrial glucocorticoid deficiency will provide a novel approach to therapy for women with HMB. The synthetic glucocorticoid dexamethasone (Dex) is a potent cortisol surrogate and glucocorticoid receptor (GR) agonist that resists 11βHSD2 inactivation. In a non-human primate study the investigators have observed a striking reduction in menstrual blood loss after Dexamethasone administration.

Objectives The investigators aim to show proof-of-concept that Dexamethasone administration in women with HMB will improve the capacity of endometrial vasculature for efficient vasoconstriction when menses commences, and hence reduce menstrual bleeding. The investigators' proposal is a novel use of an existing, well-characterised medical treatment (Dex).

Methods The Investigators propose a parallel group randomised controlled trial in women with HMB comparing Dexamethasone (over a range of potential doses) to placebo treatment. The trial design will be response-adaptive, whereby randomisation probabilities change across time to ensure that maximum information is obtained in the critical region of the underlying dose-response curve (that containing the 'optimum' dose). This has the added advantage that relatively more and more women are randomised to the doses emerging as most effective. Such a design is the most parsimonious way to enable both robust demonstration of the therapeutic effect of Dexamethasone on HMB, and reliable identification of the optimal dose to take forward for future further study in a Phase III trial.

Work Up Stage Adaptive designs such as this require a work up stage to enable the simulation modelling necessary to determine a robust final design specification with adequate power (here, the expected number of patients required lies in the range 100-108). In addition this work up stage will allow two clinical studies to be executed. Data collected in these will inform the modelling and simulation, but will also enhance mechanistic and pharmacodynamic understanding of observed Dexamethasone effect, and will be an invaluable preliminary check of safety of this 'first-in-HMB' use of oral Dexamethasone. These studies will involve treating in total 20 women with HMB with two cycles of Dexamethasone (1.5mg daily).

ELIGIBILITY:
Inclusion Criteria:

* Complaint of HMB, including women with fibroids
* Pre-menopausal
* Age 18 years and over
* Describing menstrual cycles every 21- 42 days
* Provide written informed consent prior to any study related procedures
* If of childbearing potential either agree to practice a non-hormonal method of contraception for duration of study or have a partner with a vasectomy
* Workup (Study 1 or 2)- MBL for single screening period is >= 50mL
* Adaptive Trial (Study 3)- average MBL for two screening menstrual collections is >= 50mL

Exclusion Criteria:

* Currently breast-feeding
* History or current uterus, cervix, ovarian or breast cancer
* Known severe coagulation disorder
* Glucocorticoid treatment or sex steroid administration by any route in previous 1 month
* Taking prohibited medication -
* Thyroid, renal or liver dysfunction
* Diabetes mellitus
* Treated moderate/severe hypertension
* Psychotic depressive illness
* Rare hereditary galactose intolerance, lactase deficiency or glucose galactose malabsorption (due to lactose content of trial medication)
* Has a problem with alcohol or drug abuse
* Has a mental condition rendering her unable to understand the nature and scope of the study
* Participation in treatment phase in any earlier DexFEM study (1 or 2)
* Is currently enrolled in an investigational drug or device study or participated in such a study within the previous 30 days and is still in exclusion period
* workup study 1, only, an additional exclusion criterion of any contra-indication to MRI

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Change or difference in mean laboratory measured menstrual blood loss(MBL) | 3-4months
  study1:Change in mean MBL between baseline and Dexamethasone treatment cycles. Study2:Difference in mean MBL between placebo and Dexamethasone treatment cycles.
  Study3 (adaptive):Change in mean MBL between baseline and cycles during randomised (Dexamethasone/placebo) treatment

SECONDARY OUTCOMES:
Menstrual diary score for volume of menstrual period | 3-4months
  menstrual blood loss estimated from patient's daily record of menstrual products used
Satisfaction with treatment by means of a participant completed treatment review questionnaire | 3-4months
  Participants will be asked to complete a treatment review questionnaire at the end of their study participation to elicit subjective assessment of the effect of the study treatment.
Number of participants with adverse events as a measure of safety and tolerability | 3-4months
  Participants will be asked about the occurrence of adverse events at each study visit and at each contact with the research team.Adverse events will be recorded from time of consent to 30 days after last treatment dose.
Examine effect of treatment on Period pain via participant self-report questionnaire | 3-4months
  Participants will be asked to assess levels of period pain in the menstrual diaries and in the pre and post treatment questionnaires.
Mechanistic examination of response to Dexamethasone | 2 months
  study 1 only:mechanistic variables comparing an un-treated and a treated cycle via MRI scan and endometrial biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Critchley, MBChB MD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Background] Critchley HO, Maybin JA. Molecular and cellular causes of abnormal uterine bleeding of endometrial origin. Semin Reprod Med. 2011 Sep;29(5):400-9. doi: 10.1055/s-0031-1287664. Epub 2011 Nov 7. PMID 22065326
- [Background] Rae M, Mohamad A, Price D, Hadoke PW, Walker BR, Mason JI, Hillier SG, Critchley HO. Cortisol inactivation by 11beta-hydroxysteroid dehydrogenase-2 may enhance endometrial angiogenesis via reduced thrombospondin-1 in heavy menstruation. J Clin Endocrinol Metab. 2009 Apr;94(4):1443-50. doi: 10.1210/jc.2008-1879. Epub 2009 Jan 21. PMID 19158196
- [Derived] Warner P, Whitaker LHR, Parker RA, Weir CJ, Douglas A, Hansen CH, Madhra M, Hillier SG, Saunders PTK, Iredale JP, Semple S, Slayden OD, Walker BR, Critchley HOD. Low dose dexamethasone as treatment for women with heavy menstrual bleeding: A response-adaptive randomised placebo-controlled dose-finding parallel group trial (DexFEM). EBioMedicine. 2021 Jul;69:103434. doi: 10.1016/j.ebiom.2021.103434. Epub 2021 Jul 2. PMID 34218053
- [Derived] Warner P, Weir CJ, Hansen CH, Douglas A, Madhra M, Hillier SG, Saunders PT, Iredale JP, Semple S, Walker BR, Critchley HO. Low-dose dexamethasone as a treatment for women with heavy menstrual bleeding: protocol for response-adaptive randomised placebo-controlled dose-finding parallel group trial (DexFEM). BMJ Open. 2015 Jan 14;5(1):e006837. doi: 10.1136/bmjopen-2014-006837. PMID 25588784